CLINICAL TRIAL: NCT06548256
Title: The Clinical Application of Clostridium Butyricum Miyairisan for Motor and Non-motor Symptoms in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20220001
Record Dates: First submitted 2024-05-16; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-01

CONDITIONS: Clostridium Butyricum Miyairi; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Drug: Miyarisan-BM (Clostridium Butyricum Miyairi) for 1 year, then stopped for 1 year Drug: observed for 1 year and then Miyarisan-BM (Clostridium Butyricum Miyairi) for 1 year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Miyarisan-BM (Clostridium Butyricum Miyairi) first (Experimental): Miyarisan-BM (Clostridium Butyricum Miyairi) for 1 year, then stopped for 1 year
  Interventions: Drug: Miyarisan-BM (Clostridium Butyricum Miyairi)
- Miyarisan-BM (Clostridium Butyricum Miyairi) later (Experimental): observation for 1 year and then Miyarisan-BM (Clostridium Butyricum Miyairi) for 1 year.
  Interventions: Drug: Miyarisan-BM (Clostridium Butyricum Miyairi)

INTERVENTIONS:
Drug: Miyarisan-BM (Clostridium Butyricum Miyairi) — probiotics

SUMMARY:
This is an open-label, single-center, non-randomized study to assess the efficacy of Clostridium Butyricum Miyairi on the motor and non-motor symptoms of Parkinson's disease

DETAILED DESCRIPTION:
The physician will explain the trial procedures in the outpatient, and then obtain the written informed consent to start the interview. And randomly divided into experimental and observation groups, and according to the timing of taking Miyarisan, scale evaluation and sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 20 years old, diagnosed with Parkinson's disease.

Exclusion Criteria:

* People with Parkinson's disease Dementia, or Lactose Intolerance

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 3 | 0, 3, 12, 15, 24 months
  Part 3 of this scale assesses motor performance in 33 items. Each item is scored on a scale of 0 (normal) to 4 (severe), with a total score range of 0 to 132, and higher scores mean the patient's situation is worse.
Hamilton Depression Rating Scale (HAM-D) | 0, 3, 12, 15, 24 months
  This scale assesses non-motor symptoms in 17 items, the total scale value is 50 (Scores 0 to 7 mean normal, 8 to 13 mean mild depression, 14 to 18 mean moderate depression, 19 to 22 mean severe depression, and ≥23 mean very severe depression).
Hamilton Anxiety Scale (HAM-A) | 0, 3, 12, 15, 24 months
  This scale assesses non-motor symptoms in 14 items. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where ≤17 indicates mild anxiety severity, 18-24 indicate mild to moderate anxiety severity, 25-30 indicate moderate to severe anxiety severity, >30 indicate severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical Univeristy Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No